CLINICAL TRIAL: NCT00003611
Title: Chemoprevention Trial of Acitretin Versus Placebo in Solid Organ Transplant Recipients With Multiple Prior Treated Skin Cancers
Brief Title: Acitretin in Preventing Skin Cancers in Patients With Previously Treated Skin Cancers Who Have Undergone Organ Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCCTG-969251; CDR0000066688 (Registry Identifier: PDQ (Physician Data Query)); NCI-P98-0137
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Non-melanomatous Skin Cancer
Keywords: basal cell carcinoma of the skin; squamous cell carcinoma of the skin
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Acitretin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- acitretin (Experimental): Patients receive oral acitretin daily for 2 years. Skin biopsies are obtained at 1 year from normal areas and from any areas with skin cancer for genetic studies.
  Patients are followed every 6 months.
  Interventions: Drug: acitretin
- placebo (Placebo Comparator): Patients receive placebo daily for 2 years. Skin biopsies are obtained at 1 year from normal areas and from any areas with skin cancer for genetic studies.
  Patients are followed every 6 months.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: acitretin
  Arms: acitretin
Other: placebo
  Arms: placebo

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of acitretin may be an effective way to prevent the recurrence or further development of skin cancer.

PURPOSE: Randomized clinical trial to study the effectiveness of acitretin in preventing skin cancers in patients with at least two previously treated skin cancers who have undergone organ transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the chemopreventive efficacy of acitretin in immunosuppressed solid organ transplant recipients with a history of multiple previous basal cell carcinoma (BCC) or squamous cell carcinoma (SCC) skin cancer resections.
* Evaluate human papillomavirus (HPV) as a possible etiologic cofactor in the development of cutaneous epidermal dysplasia/carcinoma from skin tissues of these patients.
* Determine the effect of acitretin on potential surrogate endpoint biomarkers and HPV DNA in normal (sun protected), sun-exposed, and dysplastic and carcinoma (SCC/BCC) skin specimens.

OUTLINE: This is a randomized study. Patients are stratified according to age (at least 18 to under 50 vs 50 to 59 vs 60 to 69 vs 70 and over), number of prior skin cancers in past 5 years (2 vs 3 vs at least 4), time since most recent skin cancer occurrence (less than 12 months vs at least 12 months), sunburn susceptibility (none vs moderate vs high), visible skin damage (mild vs moderate vs severe).

Patients receive either oral acitretin or placebo daily for 2 years. Skin biopsies are obtained at 1 year from normal areas and from any areas with skin cancer for genetic studies.

Patients are followed every 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Solid organ recipient (kidney, liver, heart, lung, or pancreas) receiving immunosuppressive agents (e.g., prednisone, other corticosteroid, azathioprine, cyclosporine, tacrolimus, mycophenolate mofetil)
* At least 6 months since transplant
* At least 2 prior (same event or separate events) basal cell carcinomas (BCC) or squamous cell carcinomas (SCC) resected

  * All visible BCC and SCC resected

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Life expectancy:

* Greater than 2 years

Hematopoietic:

* WBC at least 3400/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10.0 g/dL

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 3 times ULN
* SGOT no greater than 3 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Other:

* Not pregnant or nursing
* Fertile patients must use two effective forms of birth control for at least 1 month before, during, and at least 3 years after study
* No history of oral retinoid intolerance
* No significant, uncontrolled hyperlipidemia
* No other significant medical condition or threatened allograft rejection state where retinoid use would be contraindicated

PRIOR CONCURRENT THERAPY:

Other:

* At least 1 year since prior retinoids
* No concurrent oral vitamin A supplements, topical retinoids, or other potentially irritating skin preparations
* No alcohol during and for 2 months after study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2000-05; Primary Completion 2003-02 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
rate of new primary nonmelanoma skin cancers | Up to 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark R. Pittelkow, MD, Study Chair — Mayo Clinic
Locations (11):
- United States (11):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Health Plaza, Saint Cloud, Minnesota
  - Medcenter One Health System, Bismarck, North Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Result] Kadakia KC, Barton DL, Loprinzi CL, Sloan JA, Otley CC, Diekmann BB, Novotny PJ, Alberts SR, Limburg PJ, Pittelkow MR. Randomized controlled trial of acitretin versus placebo in patients at high-risk for basal cell or squamous cell carcinoma of the skin (North Central Cancer Treatment Group Study 969251). Cancer. 2012 Apr 15;118(8):2128-37. doi: 10.1002/cncr.26374. Epub 2011 Aug 31. PMID 21882176